CLINICAL TRIAL: NCT02429908
Title: A Prospective, Multi-Center, Post-Market Surveillance Study to Assess the Clinical Efficacy and Fusion Rates of the Zimmer TM Ardis Interbody Fusion System
Brief Title: Post-Market Surveillance Study of the TM Ardis Interbody Fusion System
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CME2013-01S
Record Dates: First submitted 2015-03-16; First posted 2015-04-29 (Estimated); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Post market study of TM-Ardis Interbody (Other): TM-Ardis TLIF MIS or Open single or multi level implant for lumbar fusion
  Interventions: Device: TM-Ardis Interbody

INTERVENTIONS:
Device: TM-Ardis Interbody — The TM Ardis implant is a single device manufactured wholly from Trabecular Metal™ (porous tantalum) material, a highly porous, three-dimensional biomaterial designed for biologic fixation. is indicated for use with autogenous bone graft as an intervertebral body fusion device at one or two contiguous levels in the lumbosacral region (L2- S1) in the treatment of degenerative disc disease (DDD) with up to Grade 1 spondylolisthesis or retrolisthesis at the involved level(s).
  Other Names: Interbody Cage

SUMMARY:
This study is a post-market clinical follow-up study to fulfill the post-market surveillance obligations according to Medical Device Directive and MEDDEV 2.12-2_Rev2_January 2012. The data collected from this study will serve the purpose of confirming safety and performance of the TM Ardis implant. The goal of this study is to demonstrate that implant is effective in reducing patient disability.

DETAILED DESCRIPTION:
This study is a post-market clinical follow-up (PMCF) study to fulfill the post-market surveillance obligations according to Medical Device Directive and MEDDEV 2.12-2_Rev2_January 2012. The data collected from this study will serve the purpose of confirming safety and performance of the TM Ardis implant. The goal of this study is to demonstrate that implant is effective in reducing patient disability, which will be assessed with the ODI questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18 years
* Degenerative disc disease DDD with up to Grade 1 spondylolisthesis or retrolis-thesis at the involved level. DDD is defined as discogenic back pain with degener-ation of the disc confirmed by history and radiographic studies.
* ODI 40 out of 100
* Back pain 4 out of 10
* Mono segmental or two level lumbosacral disease
* Skeletally mature patients
* Six months failed conservative treatment.
* Gave written consent to take part in the study by signing the Ethics Committee's approved Patient Informed Consent Form.
* Physically and mentally able to comply with the protocol, including ability to read and complete required forms and adhere to the follow-up requirements of the pro-tocol.

Exclusion Criteria:

* Prior surgical procedure at the index level(s) using the desired operative approach.
* Severe degenerative lesions at more than two level of the lumbosacral spine.
* Morbid obesity (BMI greater than or equal to 40).
* Active local infection in or near the operative region.
* Active systemic infection and/or disease.
* Severe osteoporosis or insufficient bone density, which in the medical opinion of the physician precludes surgery or contraindicates instrumentation.
* Known or suspected sensitivity to the implant materials.
* Endocrine or metabolic disorders known to affect osteogenesis (e.g.Paget's disease, renal osteodystrophy, hypothyroidism)
* Systemic disease that requires the chronic administration of nonsteroidal anti-inflammatory or steroidal drugs.
* Significant mental disorder or condition that could compromise the patient's ability to remember and comply with preoperative and postoperative instructions (e.g. current treatment for a psychiatric/psychosocial disorder, senile dementia, Alzheimer's disease, traumatic head injury)
* Neuromuscular disorder that would engender unacceptable risk of instability, implant fixation failure, or complications in postoperative care.
* Pregnant.
* Unwilling to follow postoperative instructions, in particular with respect to athletic or occupational activities.
* Current vertebral metastatic tumors.
* Symptomatic cardiac disease.
* Severe congenital or acquired vertebral deformities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-03; Primary Completion 2018-09-14 (Actual); Study Completion 2018-09-14 (Actual)

PRIMARY OUTCOMES:
Improvement in ODI score | 24 months
  mean change in score of the ODI from baseline to 24 months post surgery. A 15 point improvement in ODI score will be considered as a success.

SECONDARY OUTCOMES:
Safety - Adverse Events | 24 months
  All adverse events will be assessed by incidence and time to resolution of postoperative device-related complications and serious adverse events/ incidence and time to re-operation/ incidence and time to re-vision
Fusion rate - X-ray | 3, 6, 12 and 24 month
  will be assessed at 3, 6, 12 and 24 months with the following fusion criteria: No evidence of radiolucency surrounding more than 50% of device, translational motion <3 mm and angular motion <5°.
Patient Outcomes - Mean EQ-5D | 24 months
Modic changes - MRI | 12 and 24 months
  Modic changes will be assessed by MRI
Numerical Rating Scale (NRS) for back and leg | 3 , 6, 12, and 24 months
  Patients will grade back and leg pain with a numeric scale 0 - 10
Zung self-rating depression scale score | 3, 6, 12, & 24 months
  Patients will complete a questionaire to assess depression.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Batts, Study Director — Zimmer Biomet Spine
Locations (10):
- OLV Ziekenhuis Department Neurosurgery, Aalst, Belgium
- Canada (3):
  - Vernon Jubile Hospital, Vernon, British Columbia
  - McGill University, Montreal
  - Sunnybrook Regional Hospital, Toronto
- C.H.U. RENNES - Pontchaillou, Rennes, France
- Germany (3):
  - Klinikum Dortmund gGmbH, Dortmund
  - Asklepios Kliniken GmbH - Auguststrasse, Schwedt
  - St. Josef Hospital Troisdorf, Troisdorf
- Fundación Jiménez Díaz - Servicio de Cirugía Ortopédica y Traumatología -Avda. Reyes Católicos,, Madrid, Spain
- Sahlgrenska University Hospital Department of Orthopedics, Spine Divison, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided